CLINICAL TRIAL: NCT00748527
Title: A Cancer Research UK Randomised, Multicentre, Phase II Trial of the DNAhypomethylating Agent, 5-Aza-2'-Deoxycytidine (Decitabine) Given Intravenously in Combination With Carboplatin, Versus Carboplatin Alone Given 4 Weekly in Patients With Progressive, Advanced Ovarian Cancer
Brief Title: Carboplatin With or Without Decitabine in Treating Patients With Progressive, Advanced Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was "withdrawn" due to certain adverse events [hypersensitivity].
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CRUK-PH2/051; CDR0000613805 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2006-002324-41; MGI-CRUK-PH2/051; CTA-21106/0219/001; NCT00514124 (obsolete NCT alias)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-09

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: fallopian tube cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Decitabine

ARMS (2):
- Arm I (Active Comparator): Patients receive carboplatin IV over 30-60 minutes on day 1.
  Interventions: Drug: carboplatin
- Arm II (Experimental): Patients receive decitabine IV over 6 hours on day 1 and carboplatin IV over 30-60 minutes on day 8.
  Interventions: Drug: carboplatin; Drug: decitabine

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: decitabine — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and decitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether carboplatin is more effective with or without decitabine in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

PURPOSE: This randomized phase II trial is studying carboplatin and decitabine to see how well they work compared with carboplatin alone in treating patients with progressive, advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the response rate in patients with progressive, advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer who have methylated hMLH1 DNA in plasma treated with carboplatin with vs without decitabine.

Secondary

* To compare the response rate in all patients (regardless of methylation status) treated with these regimens.
* To compare the progression-free survival and overall survival of patients treated with these regimens.
* To compare the safety and tolerability of these regimens.
* To determine the feasibility of combining decitabine with carboplatin.
* To determine the incidence of hypersensitivity reactions to carboplatin.
* To study the relationship between peak plasma levels of decitabine and global or CpG island specific methylation.
* To study the relationship between global and gene specific methylation in peripheral blood mononuclear cells and response.

Tertiary

* To correlate the methylation status of genes associated with drug resistance detected in plasma DNA with response.
* To determine the sensitivity and specificity of methylation of genes associated with drug resistance detected in plasma DNA as a predictor of methylation status in tumor cells isolated from ascites or tumor biopsy.
* To study methylation and expression of genes in tumor cells isolated from ascites or tumor biopsy before and after treatment with decitabine and/or carboplatin.
* To investigate any correlation between methylation and expression of genes in surrogate tissues, body fluids, or tumor cells and response or progression-free survival.
* To examine markers of cell death in plasma.
* To compare the methylation in tumor taken at the time of presentation vs at the time of treatment.

OUTLINE: This is a multicenter study. Patients are stratified according to prior first-line treatment (platinum alone vs platinum and taxane vs platinum and other combination), WHO performance status (0 vs 1 vs 2), measurable disease criteria (RECIST criteria vs CA-125 criteria vs both), participating center, and the number of prior platinum-based regimens (1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carboplatin IV over 30-60 minutes on day 1.
* Arm II: Patients receive decitabine IV over 6 hours on day 1 and carboplatin IV over 30-60 minutes on day 8.

In both arms, treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for pharmacodynamic studies. Samples are assessed for methylation of hMLH1 by methylation-specific PCR; global DNA methylation by high performance liquid chromatography (HPLC) ; methylation of the MAGE-1A gene promoter by methylation-specific PCR or bisulfite pyrosequencing; and markers of apoptosis by ELISA. Pharmacokinetic studies of decitabine are also performed using blood samples from patients randomized to arm II. Ascitic fluid and/or tumor tissue samples may also be collected for pharmacodynamic studies.

After completion of study treatment, patients are followed at 28 days and then every 2 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer

  * Progressive disease as defined by RECIST criteria and/or CA-125 criteria
  * Advanced disease
* Previously treated with 1-2 prior platinum-containing regimen(s)

  * Prior hormonal therapy does not count towards the prior treatment
  * Responded to the most recent prior platinum-containing regimen(s) OR no evidence of progression during platinum-containing therapy as documented by RECIST criteria or CA-125 criteria (for patients with no macroscopic residual disease after surgery who are not evaluable by CA-125)
* Disease relapse 6-12 months after completion of the most recent platinum-containing therapy

  * Patients who received two prior lines of treatment must have had ≥ 6 months between their first and second lines of treatment
  * Patients with disease progression, as defined by CA-125 criteria alone, within 6 months after completion of their last treatment are eligible provided study treatment commences > 6 months after the last prior treatment
  * Patients with disease progression, as defined by GCIG guidelines, within 12 months after completion of their last treatment are eligible provided study treatment commences ≤ 14 months after the last prior treatment
* Measurable disease by RECIST criteria and/or CA-125 criteria

  * Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques (physical examination, CT scan, x-ray, or MRI) or as ≥ 10 mm by spiral CT scan
  * Patients with evaluable disease by CA-125 criteria are eligible provided CA-125 is ≥ 2 times upper limit of normal (ULN) within 2 weeks prior to initiating study treatment
  * Disease is not considered measurable if patient received prior mouse antibodies or if there has been medical and/or surgical interference with the peritoneum or pleura (e.g., paracentesis) within the past 28 days
* Ascites requiring therapeutic drainage allowed only if there is measurable disease by RECIST criteria

  * Ascites that do not require therapeutic drainage allowed even if disease is evaluable by CA-125 criteria alone

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Hemoglobin ≥ 10.0 g/dL
* WBC ≥ 3.0 x 10^9/L
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 30 μmol/L
* ALT and/or AST ≤ 2.5 times ULN (≤ 5 times ULN if due to tumor involvement of liver)
* EDTA/DTPA clearance ≥ 50 mL/min (uncorrected value)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 4 weeks prior to, during, and for 6 months after completion of study treatment
* No known hepatitis B, hepatitis C, or HIV positivity
* No non-malignant systemic disease, including active uncontrolled infection, that would make the patient a high medical risk
* No other current malignancies, except adequately treated cone-biopsied in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin

  * Patients who have undergone potentially curative therapy for a prior malignancy are eligible provided there is no evidence of disease for ≥ 5 years and the patient is deemed to be at low risk for recurrence
* No intolerance to carboplatin (with a dose of ≥ AUC 5), as defined by any of the following:

  * Neutropenia or thrombocytopenia causing dose delay of > 4 days on more than 2 occasions
  * Grade III or IV hypersensitivity reaction (not controlled by a desensitization regimen)
  * Hospitalization for confirmed febrile neutropenia (fever ≥ 38°C)
  * Requirement for platelet transfusion
* No other condition that, in the investigator's opinion, would not make the patient a good candidate for this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy (alopecia, grade 1 neuropathy, and certain grade 1 toxicities allowed)
* More than 28 days since prior maintenance therapy (e.g., erlotinib or bevacizumab)
* More than 4 weeks since prior radiotherapy, endocrine therapy, immunotherapy, chemotherapy, biological therapy, or investigational agents
* More than 4 weeks since prior major thoracic and/or abdominal surgery and recovered
* No other concurrent anti-cancer therapy, including radiotherapy or investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Response rate (partial response [PR] or complete response [CR]) in patients with methylated hMLH1 DNA in plasma as measured by RECIST criteria or CA-125 criteria

SECONDARY OUTCOMES:
Response rate (PR or CR) in all patients (regardless of methylation status) as measured by RECIST criteria or CA-125 criteria
Progression-free survival and overall survival
Adverse events as measured by NCI CTCAE v3.0
Total dose and dose intensity of carboplatin and decitabine
Incidence of grade 3-4 hypersensitivity reactions
Correlation between peak plasma levels of decitabine and global and CpG island specific DNA methylation in peripheral blood mononuclear cells
Correlation between response (PR or CR) and global and CpG island specific DNA methylation in peripheral blood mononuclear cells
Correlation between response (PR or CR) and CpG island specific DNA methylation in plasma DNA
CpG island specific DNA methylation in plasma and tumor DNA
CpG island specific DNA methylation in tumor DNA and expression of genes as measured by RNA or protein assays
Correlation between response (PR, CR, or stable disease) and CpG island specific DNA methylation in tumor DNA and expression of genes by RNA or protein assays
Immunoassays of proteins in plasma
CpG island specific DNA methylation in tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Stanley B. Kaye, MD, FRCP, Study Chair — Royal Marsden NHS Foundation Trust
Locations (11):
- United Kingdom (11):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Saint Bartholomew's Hospital, London, England
  - Royal Marsden - London, London, England
  - Hammersmith Hospital, London, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Royal Marsden - Surrey, Sutton, England
  - Weston General Hospital, Weston-super-Mare, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland